CLINICAL TRIAL: NCT04457518
Title: Nutritional Status in Children With Inflammatory Bowel Disease
Brief Title: Nutritional Status in Children With IBD
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Turkish Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Principal Investigator, Zarife Kuloglu, Professor, MD., Ankara University
Other Study IDs: 12.10.2011/11-7/2
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases; Child
Keywords: İnflammatory bowel disease; children; nutritional status
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition and growth retardation are major extraintestinal presentations of inflammatory bowel disease (IBD) in childhood and are especially prevalent among those with Crohn's disease. We aimed to evaluate nutritional status of children with IBD at the time of diagnosis.

DETAILED DESCRIPTION:
Data for this study will be derived from the web-based National Registry for Pediatric IBD. The children (age: ≤ 18 years) who diagnosed with IBD according to international criteria will be eligible for enrollment. Data on demographic, clinical and laboratory characteristics at the time of diagnosis were extracted from the registry. All cases in the registry will be screened for eligibility criteria by principal investigator (senior gastroenterologist). The patients with other chronic disease known affect nutritional status will be excluded. The cases who had the missing major outcome variables including symptom duration, weight, height, disease activity, disease location and phenotype at the time of diagnosis will be excluded from the analysis, if they had all of these outcome variables, they were included.

The nutritional status of participants will be evaluated based on anthropometric parameters. The weight status will be assessed by weight-for-length in children <2 years of age, and BMI-for-age in children 2 years of age and older. Height status will be evaluated by length/height-for-age in all cases. Age-and-sex specific percentile and the corresponding z score for all anthropometric parameters will be calculated in the WHOAnthro for under five years and WHOAnthroplus (WHO, Geneva, Switzerland) for those aged 5-18 years by using WHO standards and references. Z-scores between +2.0 and -2.0 for all parameters will be considered normal. Wasted/thinness and overweight will be defined by weight-for-length/BMI z score < -2.0, and > +2.0, respectively. Stunting (short stature) and tallness will be defined as length/height-for-age z score < -2.0 and > +2.0, respectively. Children will be stratified into two age groups for analysis: < 10 years of age and older. A p value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≤ 18 years
2. Diagnosis of IBD with clinical, laboratory, endoscopic and histopathologic findings
3. No other chronical diseases known affect nutritional status
4. No missing data in major variables including symptom duration, weight, height, disease activity, disease location and phenotype at the time of diagnosis

Exclusion Criteria:

1. Age: >18 years old
2. Another chronical disease known affect nutritional status
3. Missing data in major variables including symptom duration, weight, height, disease activity, disease location and phenotype at the time of diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Secondary and Tertiary Care Hospital
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
nutritional profiles of children with IBD | Day 1 of diagnosis
  evaluating nutritional profiles of children with IBD at the time of diagnosis by anthropometric parameters

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Kuloglu, M.D., Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuloglu Z, Cetin F, Urganci N, Onal Z, Sari S, Yuksekkaya H, Caltepe G, Kutluk G, Dumlupinar E; Turkish Inflammatory Bowel Disease Study Group. Nutritional characteristic of children with inflammatory bowel disease in the nationwide inflammatory bowel disease registry from the Mediterranean region. Eur J Clin Nutr. 2022 Sep;76(9):1289-1296. doi: 10.1038/s41430-022-01094-6. Epub 2022 Feb 16. PMID 35173290
- See also: Assessing and managing children at primary health-care facilities to prevent overweight and obesity in the context of the double burden of malnutrition — https://www.who.int/publications/i/item/9789241550123
- See also: Nutritional concerns in pediatric inflammatory bowel disease — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4958701/
- See also: Nutrition in Paediatric Inflammatory Bowel Disease: A Position Paper on Behalf of The Porto IBD Group of ESPGHAN — https://pubmed.ncbi.nlm.nih.gov/29570147/